CLINICAL TRIAL: NCT03330873
Title: Randomized, Controlled Trial to Assess the Efficacy of Disposable Balloon Uterine Stent and Foley Catheter in the Prevention of Adhesion Reformation After Hysteroscopic Adhesiolysis
Brief Title: The Efficacy and Safety of Disposable Balloon Uterine Stent in Patients With Asherman Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Obstetrics and Gynecology Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: No.3-20140601
Record Dates: First submitted 2017-10-18; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Intrauterine Adhesion
Keywords: Asherman syndrome; disposable balloon uterine stent; hysteroscopy; Foley catheter
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foley catheter (Experimental): After the completion of hysteroscopic adhesiolysis, Foley catheter was inserted and inflated with normal saline which was removed on the 7th day after surgery.
  Interventions: Device: Foley catheter
- Disposable balloon uterine stent (Experimental): After the completion of hysteroscopic adhesiolysis, disposable balloon uterine stent was inserted and inflated with normal saline which was removed on the 7th day after surgery.
  Interventions: Device: disposable balloon uterine stent

INTERVENTIONS:
Device: disposable balloon uterine stent — The disposable balloon uterine stent is heart-shaped that resembled the shape of the uterine cavity and could fully separate the two sides of the uterine wall and the corners of the uterus compare to Foley catheter
  Arms: Disposable balloon uterine stent
Device: Foley catheter — Foley catheter can partly separate the sides of uterus wall.
  Arms: Foley catheter

SUMMARY:
Asherman's syndrome is characterized by the presence of intrauterine adhesions (IUA) as well as symptoms such as amenorrhea, hypomenorrhea, pelvic pain, and infertility. The gold standard for the treatment of intrauterine adhesions is hysteroscopic intrauterine adhesions. The recurrence of intrauterine adhesions is a major challenge in clinical practice. The isolation of barriers in the uterine cavity may be a measure to reduce postoperative re adhesion, but the effect of different devices is different. Therefore, this study was conducted.

DETAILED DESCRIPTION:
The Foley catheter is usually inserted into the uterine after a hysteroscopic adhesiolysis and removed after on the 5-7th day after surgery. Several investigators demonstrated its favorable effect in the recurrence of adhesion after the treatment of intrauterine adhesion. Disposable balloon uterine stent is specially designed to fit into the cavity of the uterus, and usually removed on the 7th day after surgery.

ELIGIBILITY:
Inclusion Criteria:

* age 20-40 years;
* Moderate to severe intrauterine adhesion (AFS score ≥5）;
* complains of menstruation disorder and reproductive dysfunction
* Agreement to have second-look hysteroscopy
* informed consent

Exclusion Criteria:

* ovarian failure
* patients who did not proceed to second-look hysteroscopy within the specified time frame
* Contraindication of hormone

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-10-23 (Actual); Primary Completion 2018-08-20 (Estimated); Study Completion 2018-10-20 (Estimated)

PRIMARY OUTCOMES:
second diagnostic hysteroscopy | Within the first 3 months after surgery
  AFS score（The American Fertility Society classifications）

SECONDARY OUTCOMES:
Menstruation Pattern | Within the first 3 months after surgery
  Improvement or No Significant Change
Number of participants with pregnancy | one year
  Number of biochemical pregnancies and clinical pregnancies

CONTACTS AND LOCATIONS:
Overall Officials: Duan Hua, PhD, Study Chair — Beijing Obstetrics and Gynecology Hospital
Locations (1):
- Beijing Obstetrics and Gynecology Hospital，Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No